CLINICAL TRIAL: NCT05436743
Title: Efficacy of K-Y Jelly in Prevention of Postoperative Sore Throat After Nasal Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alaa Gamal (Network)
Responsible Party: Sponsor-Investigator, Alaa Gamal, Director, Egyptian Biomedical Research Network
Organization: Egyptian Biomedical Research Network (Network)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 072021
Record Dates: First submitted 2021-12-16; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Postoperative Sore Throat
MeSH Terms: interventions — K-Y jelly

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- K-Y jelly soaked packs (Experimental): K-Y jelly soaked packs inserted for pretension of postoperative sore throat
  Interventions: Drug: K-Y Jelly, Topical Gel soaked packs
- Water soaked packs (Active Comparator): Water soaked packs inserted for pretension of postoperative sore throat
  Interventions: Other: Water soaked packs

INTERVENTIONS:
Drug: K-Y Jelly, Topical Gel soaked packs — Topical Gel used as lubricant
  Arms: K-Y jelly soaked packs
Other: Water soaked packs — Water soaked packs for reduction of postoperative sore throat
  Arms: Water soaked packs

SUMMARY:
Postoperative sore throat (POST) is a fairly common side effect of general anesthesia which is caused by the mucosal injury and nerve compression associated with tracheal intubation or laryngeal mask airway device insertion. In this randomized study, the authors evaluate the effect of K-Y jelly-soaked nasopharyngeal packs on POST and postoperative nausea and vomiting in patients subjected to nasal surgery.

DETAILED DESCRIPTION:
Postoperative sore throat (POST) is a fairly common side effect of general anesthesia which is caused by the mucosal injury and nerve compression associated with tracheal intubation or laryngeal mask airway device insertion. In this randomized study, the authors evaluate the effect of K-Y jelly-soaked nasopharyngeal packs on POST and postoperative nausea and vomiting in patients subjected to nasal surgery.

The present double-blinded randomized controlled study was conducted at Al-Azhar University Hospitals, Cairo, Egypt. The study protocol was approved by the local ethical committee of Al-Azhar Faculty of Medicine and all patients provided informed consent before enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to nasal surgery under general anesthesia.

Exclusion Criteria:

* Acute of chronic nasopharyngeal conditions,
* Gastroesophageal reflux, regurgitation,
* History of postoperative sore throat,
* nasal surgery for malignant disease,
* concurrent or recent use of systemic or topical agents used for sore throat or
* Mallampati grade more than 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Postoperative sore throat | up to 6 hours postoperatively
  Postoperative sore throat

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Algarhy, Principal Investigator — Al-Azhar University
Locations (1):
- Al-Azhar University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No